CLINICAL TRIAL: NCT07265206
Title: An Exploratory Clinical Study on the Safety and Efficacy of HY001N Cell Injection in the Treatment of Relapsed or Refractory Autoimmune Neurological Diseases
Brief Title: A Study of HY001N in the Treatment of Relapsed or Refractory Neurological Autoimmune Diseases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY001N001
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Neurological Autoimmune Diseases
Keywords: CAR-T; HY001N; neurological autoimmune diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose of HY001N (Experimental)
  Interventions: Biological: HY001N cell injection

INTERVENTIONS:
Biological: HY001N cell injection — A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, HY001N.

SUMMARY:
This study is a single-arm, open-label, non-randomized clinical trial aimed at evaluating the safety, tolerability and preliminary efficacy of HY001N cell injection in the treatment of patients with relapsed/refractory Neurological Autoimmune Diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing to sign the informed consent form;
2. Aged 18-75 years, male or female;
3. At screening, subjects with relapsed/refractory antibody-mediated inflammatory neurological diseases without effective treatment, the expression of CD19+ B cells in peripheral blood and meeting the special criteria for different indications include:

   * Neuromyelitis optica spectrum disorder (NMOSD): Comply with the diagnostic criteria for NMOSD of the International panel for NMO diagnosis (IPND) in 2015 and meet the following requirements:

     1. aquaporin 4 (AQP4) -IgG positive
     2. At least one immunosuppressant has been used for more than one year and the symptoms have not been well controlled;
     3. EDSS score ≤8 points;
     4. There must be at least two relapses within 24 months prior to screening or at least one relapse within the past 12 months, and the relapses should be stable for at least 4 weeks.
   * Myasthenia gravis (MG): MG subjects who meet the MGFA classification II-IV as defined by the 2020 American Myasthenia Gravis Foundation (MGFA) diagnostic criteria and satisfy the following requirements:

     1. AChR-Ab serum positive or MuSK antibody positive;
     2. The MG-ADL score is ≥6 points, and the eye muscle score is less than 50% of the total score;
     3. There is one of the following poor control conditions in the previous treatment: i. After at least two conventional immunotherapy drugs (including hormone and non-hormone immunosuppressants) have been used for ≥1 year without treatment failure, that is, despite receiving IST treatment, ADL remains persistently impaired (persistent weakness, crisis or inability to tolerate IST); ii. At least one IST treatment has failed, and long-term PE or IVIg treatment is required to control symptoms, that is, PE or IVIg treatment for muscle weakness needs to be carried out regularly for at least two cycles in the past 12 months.
   * Chronic inflammatory demyelinating polyradiculopathy (CIDP): Meet the 2021 EAN/PNS diagnostic criteria (progressive or recurrent type), and have a corrected INCAT disability scale total score of 2-9 (with 2 points coming from leg disability), and meet the following requirements:

     1. Standardized use of at least one first-line therapy (cortisol hormone therapy, γ -globulin or plasma exchange therapy) for more than 3 months with poor symptom control;
     2. Inability to tolerate cortisol hormone, gamma globulin and plasma exchange due to side effects or other circumstances;
     3. Determined as an active disease (CIDP disease activity status [CDAS] score ≥2), (the disease must show activity and present clinically significant deterioration on at least one CIDP clinical assessment tool (including INCAT, I-RODS or mean grip strength)
   * Multiple Sclerosis (MS): According to the revised McDonald diagnostic criteria in 2017, a clinical diagnosis of MS is made, and the following three points are simultaneously met:

     a) Before ICF and in any of the following circumstances: i. Two relapses have been recorded in the past two years. ii. One recurrence was recorded within the past year. iii. The result of Gd enhanced MRI scan was positive within one year before screening. Note: If there is no positive result of Gd enhanced scan recorded in the previous year, the screening MRI scan results can be used.

     b) Neurological stability within one month before screening and baseline (including no recurrence of MS at this stage)
   * Autoimmune encephalitis (AE): According to the 2016 International Diagnostic Criteria for Autoimmune Encephalitis, the subject was diagnosed with autoimmune encephalitis and met all of the following requirements:

     1. At least one pathogenic antibody, NMDAR or LGI1, is positive;
     2. Previously standardized use of corticosteroids, at least one immunosuppressant/modulator, including CD20 monoclonal antibodies with poor symptom control or intolerance;
     3. Autoimmune encephalitis occurred within 3 months before screening;
     4. Modified Rankin Scale (mRS) score ≥2 or Clinical Assessment Scale for Autoimmune Encephalitis (CASE) score ≥4.
   * Anti-myelin oligodendrocyte glycoprotein immunoglobulin G antibody-related disease (MOGAD): Comply with the diagnostic criteria released by the International MOGAD Expert Group in 2023 and meet all of the following requirements:

     1. Serum positive for anti-MOG antibodies
     2. There was a history of ≥1 recurrence of MOGAD within 12 months prior to screening, or ≥2 episodes within 24 months prior to screening.
4. Proper organ function, complying with the following criteria :

   * Blood routine: Absolute lymphocyte count (ALC) ≥0.4×109/L, platelet count (PLT) ≥50×109/L, hemoglobin ≥80 g/L;
   * Coagulation function: International Normalized ratio (INR) ≤1.5 times the upper limit of normal (ULN), and activated partial prothrombin time (APTT) ≤1.5 times ULN;
   * Liver function: Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 times ULN, total bilirubin ≤1.5 times ULN;
   * Renal function: Serum creatinine ≤1.5×ULN or creatinine clearance rate (Cockcroft Gault formula) ≥60 mL/min;
   * Pulmonary function: Under indoor ventilation conditions, the blood oxygen saturation in the non-oxygen inhalation state is ≥92%; There is no clinically significant pleural effusion.
5. The clinical physician evaluated the patient's condition and allowed the use of glucocorticoids at a dose not exceeding 10mg of prednisone or its equivalent during the study period, and permitted the discontinuation of all immunosuppressants.
6. The subjects whose partners are fertile agree to use effective contraceptive measures throughout the treatment period and for 24 months after the treatment, and during this period, they are not allowed to donate eggs/sperm for assisted reproduction. Female subjects of childbearing age (women who have undergone sterilization surgery or have been menopausal for ≥12 months are not considered fertile) have negative urine pregnancy or blood pregnancy tests during the screening period.

Exclusion Criteria:

1. Current medical conditions or neurological disorders that may affect the effectiveness assessment, such as dementia, schizophrenia, bipolar disorder, major depressive disorder, history of multiple traumatic brain injury, current alcohol/drug abuse or dependence, or alcohol/drug dependence within the past two years.
2. Pregnancy or breastfeeding;
3. Have received organ or hematopoietic stem cell transplantation in the past;
4. There has been a history of new thrombosis or organ infarction within the past six months;
5. Patients diagnosed with active connective tissue diseases and requiring non-hormonal immunosuppressants/modulators for treatment;
6. Combined with active infections (such as sepsis, bacteremia, mycosis, uncontrolled pulmonary infection and active tuberculosis, etc.);
7. Positive for hepatitis B surface antigen (HBsAg) and/or hepatitis Be antigen (HBeAg); Positive hepatitis Be antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab), and HBV-DNA copy number greater than the measurable lower limit; Positive for hepatitis C (HCV) antibody Positive for human immunodeficiency virus (HIV) antibody; Those who test positive for syphilis (TP); The copy numbers of EBV-DNA and CMV-DNA are greater than the measurable lower limit.
8. Having undergone major surgery that was evaluated by the researcher as unsuitable for inclusion within 4 weeks prior to screening;
9. Other malignant tumors that have occurred or are currently present within the five years prior to screening are excluded, except for those with negligible risk of metastasis or death and curable tumors, such as well-treated cervical carcinoma in situ and basal cell carcinoma of the skin.
10. The patient's heart meets any of the following conditions:

    * Left ventricular ejection fraction (LVEF) ≤45%;
    * Persistent hypertension (≥160/100 MMHG) that remains uncontrolled despite standardized treatment
    * New York Heart Association (NYHA) Grade III or IV congestive heart failure or active heart disease;
    * Severe arrhythmias requiring treatment (excluding atrial fibrillation and paroxysmal supraventricular tachycardia);
    * The QTcB interval is ≥450ms for males and ≥470ms for females (QTcB=QT/RR1/2);
    * Had myocardial infarction, bypass surgery or stent surgery within 6 months prior to the study;
    * Other heart diseases that the researcher judged as unsuitable for enrollment;
11. Have received a live vaccine within 6 weeks before screening.
12. Participate in other interventional clinical studies before cell reinfusion,or receiving treatment of an active investigational drug within 5 half-lives . Those who have received active trial drug treatment, or who intend to participate in another clinical trial or receive treatment other than that stipulated in the protocol throughout the study period.
13. Those who are known to have hypersensitivity reactions to the components of the preparations used in the test;
14. Previously received CAR-T cell therapy;
15. Other conditions that the investigator considers unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) | Up to 28 days after infusion
Number of participants with adverse events (AEs)/serious adverse events (SAEs) | up to Month 36
  AEs and SAEs: The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.

SECONDARY OUTCOMES:
Number of participants with disability improvement confirmed per EDSS | up to Month 36
  NMOSD、MOGAD
Annualized relapse rate | Up to 36 months
  NMOSD、MOGAD、MS
Change from baseline in magnetic resonance imaging (MRI) metrics | up to Month 36
  NMOSD、MOGAD：MRI metrics assessed are 1) number of gadolinium-enhancing T1 lesions and 2) total number of new or enlarging hyperintense T2-weigted lesions
Number of participants with confirmed disability progression per Expanded Disability Status Scale (EDSS) | up to Month 6
  MS
Number of participants with at least 3 points improvement in Myasthenia Gravis activities of daily living (MG-ADL) score | up to Month 36
  MG
Number of participants with at least 3 point improvement in quantitative Myasthenia Gravis (QMG) score | up to Month 36
  MG
Number of participants who have obtained evidence of clinical improvement (ECI) | up to Month 36
  CIDP
Change in antibody titer | up to Month 36
Time of maximum observed blood concentration (Tmax) | up to Month 36
Maximum observed blood concentration (Cmax) | up to Month 36